CLINICAL TRIAL: NCT03319498
Title: Postpartum Urinary Retention With Essential Oils (PURE): A Randomized Control Trial of Essential Oil Vapor to Reduce Urinary Catheterization in Postpartum Women
Brief Title: Postpartum Urinary Retention With Essential Oils (PURE)
Acronym: PURE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Carmel Health System (Other)
Responsible Party: Principal Investigator, Robin Driver, Principal Investigator, Mount Carmel Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 170316-1
Record Dates: First submitted 2017-10-18; First posted 2017-10-24 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-11

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peppermint Oil Vapor (Active Comparator): Exposure of the perineum to the vapor of the active comparator, 2 ml peppermint oil. The perineum will NOT come into contact with the oil directly.
  Interventions: Other: Peppermint Oil Vapor
- Mineral Oil Vapor (Placebo Comparator): Exposure of the perineum to the vapor of the placebo comparator, 2 ml mineral oil. The perineum will NOT come into contact with the oil directly.
  Interventions: Other: Mineral Oil Vapor

INTERVENTIONS:
Other: Peppermint Oil Vapor — 2ml of the oil will be placed in the urine collection "hat" that fits into the bowl of the toilet. Participants will then sit on the toilet in normal fashion, exposing their perineum to the vapor of the oil. The perineum will NOT come into contact with the oil directly - only the vapor from the oil will contact the perineum.
  Arms: Peppermint Oil Vapor
Other: Mineral Oil Vapor — 2ml of the mineral oil will be placed in the urine collection "hat" that fits into the bowl of the toilet. Participants will then sit on the toilet in normal fashion, exposing their perineum to the vapor of the oil. The perineum will NOT come into contact with the oil directly - only the vapor from the oil will contact the perineum.
  Arms: Mineral Oil Vapor

SUMMARY:
The purpose of this study is to examine the effectiveness of peppermint oil to promote voiding and reduce urinary catheterization among postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* postpartum patients at Mount Carmel East, Mount Carmel West, and Mount Carmel St. Ann's Hospital
* 18 years or older
* able to read and understand English
* unable to spontaneously void within 6 hours after vaginal delivery or within 6 hours after straight catheter or within 6 hours after catheter removal for cesarean delivery.

Exclusion Criteria:

* patients who have an allergy to peppermint oil
* patients who have asthma
* patients who report sensitivity to smells
* patients who have a clinical condition which precludes walking/use of standard toilet

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study participants are postpartum women with urinary retention.
Enrollment: 390 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Resolution of Postpartum Urinary Retention | within 10 minutes after administering study intervention
  Spontaneous bladder voiding of at least 150 milliliters

SECONDARY OUTCOMES:
Time to resolution of urinary retention | Within 6 hours of postpartum urinary retention
  Time to resolution of postpartum urinary retention, defined as time from either 6 hours after vaginal delivery or within 6 hours after straight catheter in recovery or 6 hours after catheter removal for cesarean delivery to resolution of postpartum urinary retention.
Volume of urine voided | Within 6 hours of postpartum urinary retention
  Volume of urine voided within 10 minutes after study intervention administration, expressed in milliliters
Patient Satisfaction Level | Within one hour of study intervention administration
  defined as patient rating of "agree" or "disagree" or "don't know" to the question, "I would recommend this treatment to other patients who cannot empty their bladder after delivering a baby."

CONTACTS AND LOCATIONS:
Overall Officials: Robin L Driver, BS, Principal Investigator — Mount Carmel Health System
Locations (1):
- Mount Carmel Health System, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided